CLINICAL TRIAL: NCT06320379
Title: Evaluating Changes in Quality of Life and Digestion in Functional Dyspepsia in Adults
Brief Title: Zypan Functional Dyspepsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Ryan Bradley, Director of Research, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RB071522
Record Dates: First submitted 2023-04-03; First posted 2024-03-20 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-03

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to take either a placebo or Zypan dietary supplement three times per day for four weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zypan (Experimental)
  Interventions: Dietary Supplement: Zypan
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Zypan — The study product is a dietary supplement manufactured by Standard Process Inc (i.e., Zypan®). One serving (i.e., two tablets) contains a proprietary blend (595 mg) of the following: Betaine hydrochloride, bovine pancreas Cytosol™ extract, pepsin (1:10,000), pancreatin (3x), stearic acid (vegetable source), ammonium chloride, bovine spleen, and ovine spleen. Non active ingredients will include cellulose and calcium stearate. Participants will be instructed to take two tablets three times daily with meals
  Arms: Zypan
Dietary Supplement: Placebo Comparator — The control supplement will not contain any of the active ingredients in Zypan® and will also be manufactured by Standard Process Inc. Two tablets will contain 435 mg of cellulose (42%), 288 mg rice bran powder (28%), 201 mg of calcium lactate powder (19.5%*), 103 mg citric acid (10%), and 2.6 mg calcium stearate (0.25%)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of a readily available dietary supplement on quality of life and digestion in adults with functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* ● Adults 18-70 years of age (inclusive)

  * A self-reported history of symptoms consistent with Functional Dyspepsia (per Rome IV criteria - See Telephone Screening), and self-reported absence of organic disease and infection (e.g., Helicobacter pylori) with or without a formal diagnosis by a healthcare professional.
  * Adults ≥ 60 years of age must have had a normal upper gastrointestinal endoscopy
  * Willing to be randomized to take a daily dietary supplement or placebo over the 4-week study period
  * Not taken antibiotics or other drugs prescribed specifically for symptoms consistent with Functional Dyspepsia (per Rome IV criteria) for a period up to 1 month before the beginning of the study.
  * On a stable dose of all medications prior to study entry (i.e., consistent dose for a minimum of three months)
  * On a stable dose of dietary supplements for at least one month prior to enrollment
  * Willing to avoid initiation of new supplements and/or medications unless otherwise indicated by a healthcare professional
  * Able to communicate via email, complete computer-administered questionnaires, and to read and write in English.
  * Approved to be eligible for study participation at the discretion of the Principal Investigators, after review of the Formal Eligibility Screen results.
  * Non-smokers (including tobacco and cannabis products, combusted or vaporized)
  * Willing to provide written informed consent and to follow the required protocol

Exclusion Criteria:

* ● A self-reported history of peptic and/or duodenal ulcers, H. pylori infection, gastroesophageal reflux disease (GERD) explained by upper endoscopy, irritable bowel syndrome (IBS), and other chronic GI disorders.

  * Positive fecal occult blood test (FOBT) at the clinical screening visit
  * Current use of digestive enzyme and/or betaine HCL-containing dietary supplements
  * Current use of prescribed proton-pump inhibitors
  * Current use of drugs that interfere with gastrointestinal motility, including prokinetic agents.
  * History of previous abdominal surgery, including gastric surgery, excluding appendectomy.
  * Individuals with chronic kidney or liver disease, cancer, colorectal disease and/or other rare disorders that at the discretion of the PI or Clinical Investigator may impact their safety or confound trial results
  * Current involvement or within 14 days prior to screening of a significant diet or weight loss program (such as NutriSystem, Jenny Craig, Atkin's or other low-carb diet programs) or very low-calorie liquid diet programs (such as Optifast, Medifast, and/or HMR)
  * Hospitalization (for any reason other than a scheduled medical procedure unrelated to Functional Dyspepsia) within 3 months prior to screening
  * Malignancy within the last 5 years (with the exception of basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ of the cervix)
  * Intake of ≥ 2 standardized alcohol-containing beverages per day, 14 per week, or ≥4 in any single day within the past 14 days.
  * Individuals who do not consume, or are allergic to, animal products
  * Smoking tobacco or nicotine products (combusted or vaporized)
  * Use of illicit drugs/substances (such as but not limited to cocaine, phencyclidine (PCP), and methamphetamine) within 14 days of screening
  * Currently participating in another interventional research study, or participated in another interventional research study within 14 days of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Protein Assimilation | Baseline
  Concentrations of Amino Acids in Blood
Protein Assimilation | Week 4
  Concentrations of Amino Acids in Blood

SECONDARY OUTCOMES:
Mineral concentrations in blood | Baseline
  Mineral concentrations in blood as measured by Genova Diagnostics NutrEval
Mineral concentrations in blood | Week 4
  Mineral concentrations in blood as measured by Genova Diagnostics NutrEval
Fat-soluble vitamin concentration in blood | Baseline
  Fat-soluble vitamin concentrations in blood as measured by Genova Diagnostics NutrEval
Fat-soluble vitamins | Week 4
  Fat-soluble vitamin concentrations in blood as measured by Genova Diagnostics NutrEval
Leeds Dyspepsia Questionnaire | Baseline
  Subjective measure of digestive symptoms
Leeds Dyspepsia Questionnaire | Week 4
  Subjective measure of digestive symptoms
Patient Reported Outcomes Measurement Information System (PROMIS)-29 Physical Function Subscale | Baseline
  Subjective measure of Quality of life related to physical function
Patient Reported Outcomes Measurement Information System (PROMIS)-29 Physical Function Subscale | Week 4
  Subjective measure of Quality of life related to physical function

OTHER OUTCOMES:
Microbiota Relative Abundance and Composition | Baseline
  Objective measure of amount and types of gut microbes
Microbiota Relative Abundance and Composition | Week 4
  Objective measure of microbiota abundance, composition, diversity
Blood glucose | Baseline
  Blood concentrations of glucose
Blood glucose | Week 4
  Blood concentrations of glucose
Urea Nitrogen | Baseline
  Blood concentrations of Urea Nitrogen
Urea Nitrogen | Week 4
  Blood concentrations of Urea Nitrogen
Creatinine | Baseline
  Blood concentrations of creatinine
Creatinine | Week 4
  Blood concentrations of creatinine
Urea Nitrogen to creatinine ratio | baseline
  ratio of blood concentrations of urea nitrogen to creatinine
Urea Nitrogen to creatinine ratio | Week 4
  ratio of blood concentrations of urea nitrogen to creatinine
Sodium | Baseline
  blood concentrations of Sodium
Sodium | Week 4
  blood concentrations of Sodium
Potassium | Baseline
  blood concentrations of Potassium
Potassium | Week 4
  blood concentrations of Potassium
Chloride | Baseline
  blood concentrations of Chloride
Chloride | Week 4
  blood concentrations of Chloride
Carbon Dioxide | baseline
  blood concentration of carbon dioxide
Carbon Dioxide | week 4
  blood concentration of carbon dioxide
Calcium | Baseline
  blood concentration of calcium
Calcium | Week 4
  blood concentration of calcium
Total Protein | Baseline
  Total protein in blood
Total Protein | Week 4
  Total protein in blood
Albumin | Baseline
  Concentration of albumin in blood
Albumin | Week 4
  Concentration of albumin in blood
Globulin | baseline
  Concentration of globulin in blood
Globulin | Week 4
  Concentration of globulin in blood
Albumin to Globulin ratio | Baseline
  Ratio of the blood concentrations of albumin to globulin
Albumin to Globulin ratio | Week 4
  Ratio of the blood concentrations of albumin to globulin
Bilirubin | baseline
  Concentrations of bilirubin in blood
Bilirubin | Week 4
  Concentrations of bilirubin in blood
Alkaline Phosphatase | baseline
  Concentrations of alkaline phosphatase in blood
Alkaline Phosphatase | Week 4
  Concentrations of alkaline phosphatase in blood
aspartate aminotransferase | Baseline
  Concentrations of aspartate aminotransferase in blood
aspartate aminotransferase | Week 4
  Concentrations of aspartate aminotransferase in blood
Alanine aminotransferase | baseline
  Concentrations of Alanine aminotransferase in blood
Alanine aminotransferase | Week 4
  Concentrations of Alanine aminotransferase in blood
Estimated glomerular filtration rate | baseline
  glomerular filtration rate per 1.73 sqM estimated
Estimated glomerular filtration rate | Week 4
  glomerular filtration rate per 1.73 sqM estimated
White blood cell count | baseline
  Amount of leukocytes in blood
White blood cell count | Week 4
  Amount of leukocytes in blood
Red blood cell count | baseline
  Amount of erythrocytes in blood
Red blood cell count | Week 4
  Amount of erythrocytes in blood
Hemoglobin | baseline
  Amount of hemoglobin in blood
Hemoglobin | Week 4
  Amount of hemoglobin in blood
Hematocrit | baseline
  Amount of hematocrit in blood
Hematocrit | Week 4
  Amount of hematocrit in blood
Mean corpuscular volume | baseline
  Mean corpuscular volume of erythrocytes
Mean corpuscular volume | Week 4
  Mean corpuscular volume of erythrocytes
Mean corpuscular hemoglobin | baseline
  Mean corpuscular hemoglobin of erythrocytes
Mean corpuscular hemoglobin | Week 4
  Mean corpuscular hemoglobin of erythrocytes
Mean corpuscular hemoglobin concentration | baseline
  Mean corpuscular hemoglobin concentration of erythrocytes
Mean corpuscular hemoglobin concentration | Week 4
  Mean corpuscular hemoglobin concentration of erythrocytes
Erythrocyte distribution width | baseline
  Erythrocyte distribution width
Erythrocyte distribution width | Week 4
  Erythrocyte distribution width
Platelet count | baseline
  amount of platelets in blood
Platelet count | Week 4
  amount of platelets in blood
Neutrophils | baseline
  amount of neutrophils in blood
Neutrophils | Week 4
  amount of neutrophils in blood
Band Neutrophils | baseline
  Neutrophils band form per 100 leukocytes
Band Neutrophils | Week 4
  Neutrophils band form per 100 leukocytes
Absolute band neutrophils | baseline
  Amount of Neutrophils band form
Absolute band neutrophils | Week 4
  Amount of Neutrophils band form
Metamyelocytes | baseline
  Amount of metamyelocytes per 100 leukocytes
Metamyelocytes | Week 4
  Amount of metamyelocytes per 100 leukocytes
Absolute Metamyelocytes | baseline
  Amount of metamyelocytes
Absolute Metamyelocytes | Week 4
  Amount of metamyelocytes
Myelocytes | baseline
  Amount of metamyelocytes per 100 leukocytes
Myelocytes | Week 4
  Amount of metamyelocytes per 100 leukocytes
Absolute Myelocytes | baseline
  Amount of myelocytes
Absolute Myelocytes | Week 4
  Amount of myelocytes
Promyelocytes | baseline
  Amount of promyelocytes per 100 leukocytes
Promyelocytes | Week 4
  Amount of promyelocytes per 100 leukocytes
Absolute Promyelocytes | baseline
  Amount of promyelocytes
Absolute Promyelocytes | Week 4
  Amount of promyelocytes
Absolute Neutrophils | baseline
  Amount of neutrophils in blood
Absolute Neutrophils | Week 4
  Amount of neutrophils in blood
Lymphocytes | baseline
  Amount of lymphocytes in blood per 100 leukocytes
Lymphocytes | Week 4
  Amount of lymphocytes in blood per 100 leukocytes
Reactive Lymphocytes | baseline
  Amount of reactive lymphocytes in blood per 100 leukocytes
Reactive Lymphocytes | Week 4
  Amount of reactive lymphocytes in blood per 100 leukocytes
Absolute Lymphocytes | baseline
  Amount of reactive lymphocytes in blood
Absolute Lymphocytes | Week 4
  Amount of reactive lymphocytes in blood
Monocytes | baseline
  Amount of monocytes in blood per 100 leukocytes
Monocytes | Week 4
  Amount of monocytes in blood per 100 leukocytes
Absolute monocytes | baseline
  Amount of monocytes in blood
Absolute monocytes | Week 4
  Amount of monocytes in blood
Eosinophils | baseline
  Amount of eosinophils in blood per 100 leukocytes
Eosinophils | Week 4
  Amount of eosinophils in blood per 100 leukocytes
Absolute Eosinophils | baseline
  Amount of eosinophils in blood
Absolute Eosinophils | Week 4
  Amount of eosinophils in blood
Basophils | baseline
  Amount of basophils in blood per 100 leukocytes
Basophils | Week 4
  Amount of basophils in blood per 100 leukocytes
Absolute Basophils | baseline
  Amount of basophils in blood
Absolute Basophils | Week 4
  Amount of basophils in blood
Blasts | baseline
  Amount of blasts in blood per 100 leukocytes
Blasts | Week 4
  Amount of blasts in blood per 100 leukocytes
Absolute Blasts | baseline
  Amount of blasts in blood
Absolute Blasts | Week 4
  Amount of blasts in blood
Nucleated red blood cells | baseline
  Amount of nucleated erythrocytes per 100 leukocytes
Absolute Nucleated red blood cells | baseline
  Amount of nucleated erythrocytes in blood
Absolute Nucleated red blood cells | Week 4
  Amount of nucleated erythrocytes in blood
Platelet mean volume | baseline
  Mean volume of platelets in blood
Platelet mean volume | Week 4
  Mean volume of platelets in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Helfgott Research Institute, Portland, Oregon, United States